CLINICAL TRIAL: NCT05480761
Title: Evaluation of a 7-Day Therapeutic Trial Dose of Commercial Sucraid® (Sacrosidase) Oral Solution for Alleviating Congenital Sucrase-Isomaltase Deficiency (CSID) Symptoms in Pediatric Subjects With Low, Moderate, and Normal Sucrase Levels
Brief Title: 7-Day Trial of Sucraid for Alleviating CSID Symptoms in Subjects With Low, Moderate, and Normal Sucrase Levels
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of subject enrollment
Sponsor: QOL Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSDXP-13
Record Dates: First submitted 2022-06-28; First posted 2022-07-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2023-03

CONDITIONS: Congenital Sucrase-Isomaltase Deficiency; CSID; Sucrase Isomaltase Deficiency
Keywords: www.tummyachestudy.com
MeSH Terms: conditions — Sucrase-isomaltase deficiency, congenital | interventions — beta-Fructofuranosidase; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Open Labeled Commercial Sucraid (Experimental): All subjects will complete a 7-day treatment period of open-labeled FDA approved commercial Sucraid.
  Interventions: Biological: Sucraid (sacrosidase) Oral Solution 8500 IU/mL

INTERVENTIONS:
Biological: Sucraid (sacrosidase) Oral Solution 8500 IU/mL — Sucraid is a pale yellow to colorless, clear solution of glycerol, water, and citric acid, with a pleasant, sweet taste. Each milliliter of Sucraid contains 8,500 IU of the enzyme sacrosidase, the active ingredient.
  Other Names: Sucraid; Sacrosidase

SUMMARY:
This is a Phase 4, U.S. only, multi-center study using a 7-day therapeutic response dose (TRD) of commercial Sucraid® to assess the response of treatment in 1100 symptomatic pediatric (6 months to 17 years old) subjects with low, moderate, and normal sucrase activity determined by a disaccharidase assay via EGD within 1 year of the Screening Visit. This study will also explore the relationship between known genetic CSID mutations and sucrase activities via (EGD) disaccharidase assay (low, moderate, and normal).

DETAILED DESCRIPTION:
This phase 4 study will evaluate the response to Sucraid® in pediatric subjects aged 6 months to 17 years old with low (< 25 µM/min/gram protein), moderate (25-35 µM/min/gram protein), and normal (> 55 µM/min/gram protein) sucrase activities. Subjects with a sucrase level via disaccharidase assay from an EGD within 1 year of informed consent/assent, a normal histological interpretation, and at the discretion of the investigator, at least one symptom of carbohydrate maldigestion (CMS) of postprandial diarrhea, abdominal pain, gas/bloating, or defecation urgency at least 3 times per week for the past 3 months or more will be eligible for study participation. This study will also explore the relationship between three groups of sucrase levels from the EGD disaccharidase assay and the genetic test. This study will consist of a Screening Visit, Run-in Period, Baseline Visit, Treatment Period, and Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with documented disaccharidase assay levels of lactase, sucrase, maltase, and palatinase via EGD disaccharidase assay (DA) performed no more than 1 year prior to enrollment with normal histological interpretation. Eligible subjects will be enrolled into the following study groups based on their documented sucrase level.
* DA Sucrase < 25 (n=500)
* DA Sucrase 25-35 (n=500)
* DA Sucrase >55 (n=100)
* At the discretion of the investigator, subject is suspected of CSID and has at least one symptom of diarrhea, abdominal pain, gas/bloating, nausea, or borborygmi at least 3x per week for the past 3 months or more.
* Subject or parent/guardian must provide informed consent/assent prior to any study procedures being performed.
* Subject is a U.S. resident.
* Subject is male or female, ages 6 months to 17 years old.
* Subject/parent or guardian is willing and able to complete necessary study procedures including following study instructions, completing electronic questionnaires via a personal mobile device, attending study visits and, in the Investigator's judgment, is sufficiently stable to participate in the study.
* Subject/ parent or guardian must be able to read or understand the English language.
* Subject or parent/guardian must have their own Android or Apple device for BYOD.

Exclusion Criteria:

* Females who are lactating or pregnant.
* Subjects with allergy to sucrose, yeast, papain, or glycerol.
* Subjects with causes of abdominal pain or altered bowel habits other than CSID such as inflammatory bowel disease, celiac disease, eosinophilic gastrointestinal disorder, pancreatitis, or gastrointestinal bleeding.
* Subjects with a history of diabetes mellitus.
* Subjects with a recent febrile illness (5 days prior to study).
* Subjects that do not have the mental capacity to understand the study requirements and are unable to comply.
* Subject has major physical or psychiatric illness within the last 6 months that in the opinion of the investigator would affect the subject's ability to complete the trial.
* Subject has previously used Sucraid®.
* Subject has uncontrolled systematic disease.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Effects of Sucraid® treatment on gastrointestinal symptoms in subjects with low, moderate, and normal disaccharidase assay sucrase levels from an esophagogastroduodenoscopy (EGD). | Post 7-day run-in period plus 7-day treatment period.
  The primary endpoint will be the difference observed between the average symptom severity/frequency score during the 7-day treatment period and the 7-day run-in period as determined by the Daily Symptom Questionnaire using a scale from 0 to 5 or more.

SECONDARY OUTCOMES:
Explore the relationship between known genetic CSID mutations and sucrase activities via (EGD) disaccharidase assay (low, moderate, and normal). | Up to 2 years
  The number and percentage of subjects with genetic CSID mutations will also be examined in low, moderate, and normal sucrase study group.

CONTACTS AND LOCATIONS:
Overall Officials: Weng Tao, M.D., Ph. D, Principal Investigator — QOL Medical
Locations (20):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kidz Medical, Coral Gables, Florida
  - Orlando Health, Orlando, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Center for Digestive Health Care, LLC, Atlanta, Georgia
  - University of Maryland Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - GI Associates, Flowood, Mississippi
  - Happy Tummies, Flowood, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Atlantic Health System, Morristown, New Jersey
  - WNY Pediatric Gastroenterology, Buffalo, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Measurable Outcomes Research, Oklahoma City, Oklahoma
  - Prisma Health, Greenville, South Carolina
  - GI For Kids, PLLC, Knoxville, Tennessee
  - Newco 3A Research,LLC DBA 3A Research, El Paso, Texas
  - Pediatric GI of El Paso, LLC, El Paso, Texas
  - McGovern Medical School of UT Health, Houston, Texas